CLINICAL TRIAL: NCT05838222
Title: Implementation and Efficacy of Solution Focused Interventions Within an Integrated Behavioral Health Setting
Brief Title: Integrating Solution Focused Interventions in Integrated Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Orion Mowbray, Associate Dean of Research, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00006727
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Depression; Diabetes Mellitus; Hypertension; Anxiety Disorders
Keywords: Integrated care; Solution focused; Primary Care; co occurring disorders
MeSH Terms: conditions — Depression; Diabetes Mellitus; Hypertension; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Pretest-posttest experimental design with a treatment as usual group and an intervention group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive 3 sessions of SFBT from a licensed therapist in addition to treatment as usual
  Interventions: Behavioral: Solution Focused Intervention; Other: Treatment as Usual
- Control (Active Comparator): This group will be the treatment as usual group who will receive primary care treatment without the SFBT intervention
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Solution Focused Intervention — A short term, goal focused, therapeutic approach which helps patients address problems contributing to health and mental health challenges
  Arms: Intervention Group
Other: Treatment as Usual — The patient receives standardized care from primary care team without the SFBT intervention

SUMMARY:
Integrated behavioral healthcare (IBH) emerged to address the high prevalence of psychosocial issues endemic to primary care settings coupled with primary care provider's discomfort in addressing psychosocial issues. IBH addresses the lack of psychosocial care in primary care settings by expanding the traditional healthcare team through the inclusion of a behavioral health provider (clinical social worker, licensed psychologist, etc.). The behavioral health provider utilizes evidenced based interventions to support the healthcare team with addressing a wide range of healthcare concerns. Solution Focused Brief Therapy (SFBT) provides a promising treatment approach within IBH settings due to the high productivity standards within primary care and the efficient, solution based style foundational to SFBT. In addition, SFBT is strengths based and emphasizes patient centered approaches which primary care aspires to achieve. Despite the natural fit, there is a paucity of research regarding SFBT within integrated care settings in general, and for specific disease states. The purpose of this study is to assess the efficacy of SFBT within an IBH setting in the treatment of depression while assessing for commensurate improvement with traditional healthcare markers such as A1C, blood pressure, pulse, and weight. In addition, scaling questions will be utilized to assess for increase in core SFBT constructs to include self-awareness of strengths, future hope, and increased ability to problem solve. A pre-posttest experimental design will assess the differences between those receiving SFBT and treatment as usual across symptoms of depression, SFBT core attributes, and health outcomes.

DETAILED DESCRIPTION:
Integrated behavioral healthcare (IBH) emerged to address the high prevalence of psychosocial issues endemic to primary care settings coupled with primary care provider's discomfort in addressing psychosocial issue. IBH addresses the lack of psychosocial care in primary care settings by expanding the traditional healthcare team through the inclusion of a behavioral health provider (clinical social worker, licensed psychologist, etc.). The behavioral health provider utilizes evidenced based interventions to support the healthcare team with addressing a wide range of healthcare concerns. Solution Focused Brief Therapy (SFBT) provides a promising treatment approach within IBH settings due to the high productivity standards within primary care and the efficient, solution based style foundational to SFBT. In addition, SFBT is strengths based and emphasizes patient centered approaches which primary care aspires to achieve. Despite the natural fit, there is a paucity of research regarding SFBT within integrated care settings in general, and for specific disease states. The purpose of this study is to assess the efficacy of SFBT within an IBH setting in the treatment of depression while assessing for commensurate improvement with traditional healthcare markers such as A1C, blood pressure, pulse, and weight. In addition, scaling questions will be utilized to assess for increase in core SFBT constructs to include self-awareness of strengths, future hope, and increased ability to problem solve. A pre-posttest experimental design will assess the differences between those receiving SFBT and treatment as usual across symptoms of depression, SFBT core attributes, and health outcomes.

Study Aims

The purpose of this study is to examine the efficacy of SFBT in an integrated care setting for addressing depressive symptoms and health outcomes among patients with depression. The study aims are to:

Aim 1: Assess SFBT's impact on core SFBT constructs (hope, connection with important people, strengths). Measure SFBT constructs in both the control and treatment group and assess differences between the two groups

Aim 2: Assess efficacy of SFBT for depression. Examine differences between the treatment and control group for depression scores utilizing the PHQ-9.

Aim 3: Assess efficacy of treating co occurring healthcare conditions. Key outcomes of blood pressure control and HbA1c will be compared for those who have a co-occurring chronic illness such as diabetes or hypertension.

Aim 4: Evaluate implementation measures such as fidelity, acceptance, and feasibility with both patients and healthcare staff.

Method

Sample and procedure The proposed research will use a pretest-posttest experimental design where the intervention group will receive a standardized integrated care treatment protocol along with SFBT. The control group will only receive a standardized integrated care treatment protocol; in this setting access to primary care and potential referral to co located treatment. Based on an existing partnership with the Principal Investigator, participants will be recruited from a primary care clinic in the state of Georgia. Patients who have scored at or above 10 on the PHQ-9 will be considered as eligible to participate in the study. After intake and initial depression screening, any patients who have scored at or above 10 on the PHQ-9 will be considered as eligible to participate in the study. Following the consent process, participants will be randomly assigned using a random number generator process to either the SFBT treatment condition or treatment as usual condition. Individuals in the SFBT condition will receive standard integrated care protocol, plus three sessions of SFBT. The control group will only receive the standard integrated care protocol from a primary care provider. A minimum of 50 participants will be recruited into this study. A power analysis using the software G*Power shows that a sample of 48 participants will adequately power all statistical testing processes and permit the detection of medium to small effects (d = .20), given the design of the research. To ensure effective delivery of SFBT, the co-investigator will be enrolled in a Solution Focused Online Intensive Training program provided by The Institute for Solution Focused Therapy to gain a robust foundational understanding of SFBT and to ensure fidelity of the provision of SFBT within the research process. The training is online, asynchronous and uses readings, lectures, and mock interviews with patients; participants are also tested on their knowledge via online test at the end of each module. In addition, a SFBT fidelity scale will also be used to ensure service delivery is consistent SFBT best practices. The scale will be utilized by the clinician as a self-assessment to ensure SFBT fidelity.

Measures The dependent variables within the study will be 1) Symptoms of depression, 2) SFBT attributes, 3) Health outcomes, and 4) key implementation measures. Additional demographic measures will also be examined as potential control or moderating variables. The independent variable within the study will be the receipt of SFBT or treatment as usual (TAU).

Symptoms of depression. Depression will be measured at both pretest and posttest with the PHQ-9. The PHQ-9 is a standard assessment utilized in all federally qualified health centers and many primary care clinics and is therefore already embedded in the clinic workflow. The PHQ-9 has an established history of predictive validity and acceptable sensitivity (88%) and specificity (88%).

SFBT attributes. These will be assessed at both pretest and posttest with scaled questions including hope, patient strengths, and connection to important people.

Health outcomes. These outcomes will be assessed through patient chart review at both pretest and posttest. These measures will include traditional healthcare markers such as blood pressure, weight, pulse, and A1C measurements.

Demographic measures. These measures will be collected only at baseline and will include age, gender, race, ethnicity, sexual orientation, education, income, and marital status.

Implementation variables: Feasibility, Acceptability, and Appropriateness. The Acceptability of Intervention Measure (AIM), Feasibility of Intervention Measure (FIM), and Intervention Appropriateness Measure (IAM) will be provided to both patients and providers at baseline and at the end of study to determine their perception of the intervention within the primary care setting .

Data analysis plan To assess the utilization and efficacy of SFBT within an integrated care setting, participants who receive SFBT will be compared to those who receive TAU. Given the experimental nature of the research design, a factorial design ANOVA will be utilized to examine changes within each group (SFBT vs. TAU) from pretest to posttest, and changes between groups (SFT vs. TAU) at pretest or posttest. Demographic measures will be examined to ensure adequate randomization between groups, as well as for their role in potential within-group effects associated with identified outcomes. All analyses will be completed using the statistical software packages of SAS.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* PHQ9>10

Exclusion Criteria:

* No significant co occurring mental health disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Solution Focused Scaling Questions | 4 months
  The authors utilized a solution-focused treatment manual to extract the essential ingredients of solution-focused treatment and create a scale measuring the degree to which participants 1) have experienced hope, 2) experienced connection to important people, 3) identified their strengths, 4) have hope for a "good" future, and 5) believe they could solve problems in their lives over the past two weeks. Each of these questions occurred on a 1-10 scale where 1 was "not at all" and 10 was "completely." This screening tool was provided to participants in paper format where participants self-administered the survey.
Depression outcomes | 4 months
  Assess efficacy of SFBT for depression. The investigator will examine differences between the treatment and control group for depression scores utilizing the patient health questionnaire (PHQ-9.)
Diabetes Outcomes | 4 months
  Assess efficacy of SFBT for diabetes. The investigator will examine differences between the treatment and control group for depression scores utilizing HbA1c.
Acceptability measure | 4 months
  Evaluate acceptability for SFBT. The Acceptability of Intervention measure (AIM) will be used to assess the acceptability of the intervention for the treatment group. The AIM measures acceptability by asking participants whether the intervention 1) met their approval, 2) is appealing to them, 3) whether they like the intervention, and 4) whether they would welcome the intervention. A 5-point Likert scale is utilized to assess each of these domains. The scale will be self-administered by participants.
Feasibility measure | 4 months
  Evaluate feasibility for SFBT. The Feasibility of Intervention measure (FIM) will be used to assess the feasibility of the intervention for the treatment group. The FIM assesses whether the participant believes that the intervention seems 1) implementable, 2) possible, 3) doable, and 4) easy to use. A 5-point Likert scale is utilized to assess each of these domains. The scale will be self-administered by participants.

SECONDARY OUTCOMES:
Hypertension | 4 months
  Assess efficacy of SFBT for hypertension. The investigator will examine differences between the treatment and control group for depression scores utilizing blood pressure readings.

CONTACTS AND LOCATIONS:
Overall Officials: Orion Mowbray, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooper ZW, Johnson L. Strategies for Fidelity Monitoring a Solution-Focused Brief Intervention in a Randomized Clinical Trial. J Clin Psychol Med Settings. 2025 Sep;32(3):421-430. doi: 10.1007/s10880-025-10063-7. Epub 2025 Jan 28. PMID 39873935
- [Derived] Cooper ZW, Mowbray O, Ali MK, Johnson LCM. Addressing depression and comorbid health conditions through solution-focused brief therapy in an integrated care setting: a randomized clinical trial. BMC Prim Care. 2024 Aug 23;25(1):313. doi: 10.1186/s12875-024-02561-8. PMID 39179982